CLINICAL TRIAL: NCT01280734
Title: Randomised, Double-blind, 3-way Crossover, Single Dose, Placebo-controlled Study Investigating the Effect on Postural Instability of Melatonin and Zolpidem in Healthy Adult Subjects Aged of 55 to 64 Years.
Brief Title: Investigation of Melatonin and Zolpidem Effect on Postural Instability in Healthy Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Neurim-PIS1; 2010-023745-29 (EudraCT Number)
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Postural Instability
Keywords: melatonin; circadin; zolpidem; body sway; postural instability
MeSH Terms: interventions — Melatonin; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melatonin (Active Comparator): Circadin(R) 2 mg tablet 2 hours at 23:00
  Interventions: Drug: Circadin (R) 2 mg
- Zolpidem (Active Comparator): Stilnox (R) 10 mg tablet at 23:00
  Interventions: Drug: Stilnox (R) 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Circadin (R) 2 mg — One 2 mg tablet at 23:00
  Arms: Melatonin
Drug: Stilnox (R) 10 mg — One 10 mg encapsulated tablet at 23:00
  Arms: Zolpidem
Drug: Placebo — One tablet or encapsulated tablet at 23:00
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, 3-way crossover, single dose, placebo-controlled study investigating the effect on night time awakening body sway of melatonin and zolpidem in healthy adult subjects aged of 55 to 64 years.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have signed an informed consent form.
2. The subject is a healthy man or woman. Women of child bearing potential or within two years of menopause must have negative urine pregnancy test at screening and use contraceptives as indicated in the protocol.
3. The subject is 55 to 64 years of age (extremes included).
4. The subject has a BMI >19 kg/m2 and < 30 kg/m2 at the Screening Visit.
5. The subject has a normal circadian rhythm, defined as a person who usually wakes between 06:00 and 09:00 and goes to sleep between 21:00 and 24:00.
6. The subject is, in the opinion of the investigator, generally healthy based on assessment of medical history and examination at screening
7. The subject is affiliated with, or beneficiary of a social security system.

Major Exclusion Criteria:

1. The subject has taken disallowed medication within 1 week prior to the first dose of IMP (or within 5 half-lives prior to admission for any medication ingested, whichever is longer). Disallowed medication is any prescribed medication or over-the-counter (OTC) medication as well as any herbal medicine known to interfere with the metabolic CYP pathways, such as St. John's Wort (except for hormonal contraceptives or hormonal substitution therapy). Subjects who have taken any non-prescribed systemic or topical medication may still be entered into the study if, in the opinion of the investigator, the medication will not interfere with the study procedures, study results, or compromise safety.
2. The subject weighs >136 kg.
3. The subject cannot stand erect and unsupported for more than 2 to 3 minutes or loses balance when standing on a fixed surface with eyes opened.
4. The subject has an excessive consumption of beverages on xanthine bases (more than 4 cups or glasses daily).
5. The subject has a presence or history of alcohol abuse defined as alcohol consumption greater than 21 units per week for men and greater than 14 units per week for women; or a presence or history of drug abuse within the last 6 months, or a history of substance abuse deemed relevant by the investigator.
6. The subject has taken any investigational products including these IMPs (zolpidem, melatonin) within 3 months prior to admission on Day 1.
7. The subject has taken these IMPs earlier in this clinical study.
8. The subject has known hypersensitivity to the melatonin, zolpidem or their excipients.
9. The subject has a history of severe drug allergy or hypersensitivity.
10. The subject is pregnant or breastfeeding.
11. The subject has a presence or history of sleep disorder, fainting, cardiovascular diseases, carotid sinus syndrome, relevant dizziness or arrhythmia.
12. The subject has a history of or presence of any clinically relevant immunological, cardiovascular, pulmonary, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, systemic, ocular or psychiatric or infectious disease or other major disorder, or sign of acute illness.
13. The subject has a history of cancer, other than basal cell or Stage 1 squamous cell carcinoma of the skin, which has not been in remission for at least 5 years before the first dose of IMP.

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Body sway | 4 hours post IMP adminstration

SECONDARY OUTCOMES:
Body Sway | 1.5 hours post administration

CONTACTS AND LOCATIONS:
Locations (1):
- Forenap, Rouffach, France